CLINICAL TRIAL: NCT01477463
Title: Pilot Trial to Evaluate the Effect of Vitamin D on Melanocyte Biomarkers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Jean Yuh Tang, Associate Professor of Dermatology, Stanford University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: SKIN0010; SU-10272011-8570 (Other: Stanford University); IRB-22207 (Other: Stanford University); 5K23AR056736 (NIH)
Record Dates: First submitted 2011-11-17; First posted 2011-11-22 (Estimated); Results first posted 2016-12-23 (Estimated); Last update posted 2016-12-23 (Estimated); Status verified 2016-10

CONDITIONS: Melanoma, Skin
Keywords: quality of life
MeSH Terms: conditions — Melanoma | interventions — Cholecalciferol; 25-hydroxyvitamin D3-3-(1,2-epoxypropyl)ether; Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: Vitamin D (Experimental): 4,000 IU oral vitamin D3
  Interventions: Drug: Vitamin D3
- Arm B: Placebo + Vitamin D (Experimental): Placebo + 4000 IU oral Vitamin D3
  Interventions: Drug: placebo and vitamin D

INTERVENTIONS:
Drug: Vitamin D3 — 4,000 IU oral vitamin D3
  Other Names: 25-hydroxy D3
  Arms: Arm A: Vitamin D
Drug: placebo and vitamin D
  Other Names: inactive tablet and 25-hydroxy D3
  Arms: Arm B: Placebo + Vitamin D

SUMMARY:
The purpose of this study is to determine the signaling pathways and changes in gene expression in melanocytes of subjects with a history of non-melanoma skin cancer who are exposed to oral vitamin D. If vitamin D is found to inhibit a signaling pathway involved in the development of melanoma such as BRAF, a protein involved in cell proliferation, then oral vitamin D could be explored further as a chemoprevention for melanoma skin cancer.

DETAILED DESCRIPTION:
Background:

Vitamin D is an important hormone that has multiple genetic effects in different tissue types that are mediated by signaling through the vitamin D receptor.

Recent studies have shown that vitamin D signaling results in decreased innate immunity and increased adaptive immunity.

Multiple epidemiologic studies have suggested that vitamin D may play a role in decreasing the risk of developing multiple types of cancer, including skin cancer.

In the context of the relative success of novel immune-related therapies including PD1 inhibitors, which improves immuno-surveillance, and ipilimumab, which suppresses T cell response, there is increased promise for treatment strategies that activate innate immunity. This led us to ask the question of whether vitamin D could increase immune surveillance for melanoma via increased activity of the adaptive immune system.

Prior studies performed by our group and others have suggested that vitamin D may play a role in decreasing melanoma risk. An epidemiologic study from the Women's Health Initiative showed that women with a prior history of NMSC who received calcium and vitamin D supplementation had a lower risk of subsequently developing melanoma. At the same time, women with a lower serum vitamin D level had a higher risk of developing melanoma. Furthermore, a recent clinical study showed that vitamin D supplementation increases serum vitamin D levels and ultimately results in increased vitamin D receptor signaling in benign nevi.

Taken together, this findings led us to ask whether oral vitamin D supplementation could impact immune signaling in benign nevi and potentially underpin a theoretical chemo-preventive role for vitamin D in melanoma.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 - 75
2. Female
3. White race/ethnicity
4. With history of non-melanoma skin cancer
5. Has 12-16 moles upon skin examination
6. Consents to 6-12 moles biopsies over 2-3 clinic visits (2-4 months)
7. Consents to ingesting oral vitamin D3 or placebo daily for 2-4 months
8. Consents to abstaining from other multivitamins during study
9. Consents to research use of their tissue and blood samples
10. Agrees to apply a sunscreen of SPF 45 during study -

Exclusion Criteria:

1. History or current evidence of hyperparathyroidism, hypercalcemia, renal calculi, or other renal disease.
2. History or current evidence of malabsorptive illnesses, such as IBD, or liver disease that would impair uptake or metabolism of vitamin D.
3. History or current evidence of hyperthyroidism that would increase metabolism of vitamin D.
4. History or current evidence of immunosuppression (cancer, autoimmune disease) or taking immunosuppressive drugs.
5. Currently taking medications that would affect metabolism of vitamin D (anticonvulsants, corticosteroids, H2-receptor antagonists).
6. Currently taking medications that predispose to hypercalcemia (digoxin, lithium, thiazide diuretics) or other electrolyte disturbances (aluminum hydroxide)
7. Pregnancy

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-09; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean Y Tang, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University Cancer Institute, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Results will be submitted to scientific journal for publication.

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm B: Placebo: Placebo - patients may cross over to vitamin D3 treatment after placebo treatment
Period: Overall Study
Arm/Group | Arm A: Vitamin D | Arm B: Placebo
Started | 18 | 6
Completed | 18 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm B: Placebo: Placebo - subjects may cross over to vitamin D treatment after placebo treatment is complete
- Total: Total of all reporting groups
Arm/Group | Arm A: Vitamin D | Arm B: Placebo | Total
Number analyzed (Participants) | 18 | 6 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.2 (12.6) | 55.8 (5.7) | 56.1 (10.6)
Gender [Count of Participants; unit: Participants]
  Female | 18 | 6 | 24
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 18 | 6 | 24

OUTCOME MEASURES:

1. Primary Outcome: Number of Genes That Showed Changes in Expression After Vitamin D Treatment
Description: Normal cells have a complex series of molecular signals that allow communication between cells and to the cell nucleus. These signals work together to control one or more cell functions, such as cell division or cell death. Abnormal signaling activity caused by changes in gene expression can lead to cancer. An understanding of abnormal signaling, both in the tumor and in normal tissues, may lead to new therapies in cancer patients. We wish to identify changes in molecular signaling that occur in the development of melanoma that might be suppressed in benign nevi (moles) in response to vitamin D supplementation.
Time Frame: 2 years
Population: All subjects treated with vitamin D3.
Measure: Number; unit: number of genes
Groups:
- All Patients Treated With Vitamin D3: 4,000 IU oral vitamin D3
  Vitamin D3: 4,000 IU oral vitamin D3
Arm/Group | All Patients Treated With Vitamin D3
Number analyzed (Participants) | 18
number of genes | 270

2. Primary Outcome: Number of Genes Differentialy Regulated in Melanoma That Showed Changes in Expression After Vitamin D Treatment
Description: We utilized a prior gene expression study that compared malignant melanoma cells to benign nevi (moles) and identified over 2300 genes that were differentially regulated in melanoma compared to benign nevi. There were approximately 270 genes in our data set that showed changes in expression after vitamin D treatment. We wish to identify overlap between these two groups.
Time Frame: 2 years
Measure: Number; unit: number of genes
Arm/Group | All Patients Treated With Vitamin D3
Number analyzed (Participants) | 18
number of genes | 47

3. Secondary Outcome: Vitamin D Toxicity
Description: serum 25(OH)D for
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: ng/ml
Groups:
- Arm B: Placebo: Placebo (inactive capsule)
Arm/Group | Arm A: Vitamin D | Arm B: Placebo
Number analyzed (Participants) | 18 | 6
ng/ml | 47.11 (14.5) | 29.83 (4.02)

4. Secondary Outcome: Incidence of Hypercalcemia for Vitamin D Toxicity
Description: Calcium levels
Time Frame: 2 years
Measure: Number; unit: participants
Groups:
- Arm B: Placebo: Placebo - inactive capsule
Arm/Group | Arm A: Vitamin D | Arm B: Placebo
Number analyzed (Participants) | 18 | 6
participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | Arm A: Vitamin D | Arm B: Placebo
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/6
Other Adverse Events (participants affected / at risk) | 0/18 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No